CLINICAL TRIAL: NCT01063764
Title: An Open Label, Single-Arm, Multi-Center Study on the Efficacy, Safety and Pharmacokinetics of Levetiracetam in Pediatric Patients (4 to 16 Years) With Partial Seizures Despite Treatment With 1 or 2 Anti-Epileptic Drugs
Brief Title: An Open Label Study of Levetiracetam in Japanese Pediatric Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01223; 2014-004335-39 (EudraCT Number)
Record Dates: First submitted 2010-02-01; First posted 2010-02-05 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy; Partial Seizures
Keywords: Keppra; Levetiracetam; Children; Epilepsy; Partial Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Open-label, single-arm
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — First Period: Dry syrup 50 %, 20 mg/kg/day or 1000 mg/day, 40 mg/kg/day or 2000 mg/day, 60 mg/kg/day or 3000 mg/day, twice daily administration Per Os (PO) for 14 weeks.
  Second Period: Dry syrup 50 % or tablets (250 mg and 500 mg strengths), 20 to 60 mg/kg/day or 1000 to 3000 mg/day, twice daily administration Per Os (PO) until indication granted.
  Other Names: Keppra

SUMMARY:
Objective of the First Period: To evaluate the efficacy of Levetiracetam dry syrup at doses up to a maximum of 60 mg/kg/day or 3000 mg/day used as an adjunctive therapy in Japanese pediatric patients (4 to 16 years) with uncontrolled partial seizures despite treatment with 1 or 2 anti-epileptic drug(s).

DETAILED DESCRIPTION:
Objectives of the Second Period: To provide the Levetiracetam treatment to subjects who are judged by the investigators to benefit from the long-term treatment and who are willing to continuously receive this drug. To continuously evaluate the safety of the Levetiracetam long-term administration at doses ranging from 20 mg/kg/day or 1000 mg/day to 60 mg/kg/day or 3000 mg/day in subjects who completed the First Period of this study.

ELIGIBILITY:
Inclusion Criteria:

* The patient has partial Epilepsy and the diagnosis must be confirmed in the last 6 months
* The patients must be on a stable 1 or 2 anti-epileptic drug(s) treatment during the 4 weeks prior to Baseline and must have at least 8 partial seizures during the 8-week prospective Baseline Period
* Patient at the age of 4 to 16 years, and at the body weight of 11 to 82 kg

Exclusion Criteria:

* The patient has a treatable seizure etiology
* The patient has Epilepsy secondary to a progressive cerebral disease or any other progressively neurodegenerative disease, including Rasmussen and Landau-Kleffner diseases
* The patient has a history of status Epilepticus during the 3 months prior to Visit 1
* The patient has a past and present history of pseudo seizures
* The patient has a current diagnosis of Lennox-Gastaut syndrome

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (29):
- Japan (29):
  - 21, Chūō
  - 12, Hakodate
  - 22, Hamamatsu
  - 28, Hiroshima
  - 7, Izumi
  - 9, Kobe
  - 3, Kodaira
  - 30, Koga
  - 10, Kōshi
  - 31, Kurume
  - 23, Kyoto
  - 2, Nagaoka
  - 5, Nagoya
  - 6, Nagoya
  - 8, Neyagawa
  - 1, Niigata
  - 27, Okayama
  - 24, Osaka
  - 25, Osaka
  - 11, Sapporo
  - 13, Sendai
  - 4, Shizuoka
  - 26, Takatsuki
  - 16, Tokyo
  - 17, Tokyo
  - 15, Yachiyo
  - 14, Yamagata
  - 19, Yokohama
  - 20, Yokohama

REFERENCES:
- [Result] Nakamura H, Osawa M, Yokoyama T, Yoshida K, Suzuki A. [Efficacy and safety of levetiracetam as adjunctive therapy in Japanese children with uncontrolled partial-onset seizures: multicenter and open-label study (N01223), short term evaluation]. Brain Nerve. 2013 Sep;65(9):1083-92. Japanese. PMID 24018745
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Full Analysis Set (FAS) includes all subjects taking at least one dose of study medication. Per-Protocol Set (PPS) is a subset of the FAS, consisting of subjects without major protocol violations affecting the primary efficacy variable.
Pre-assignment Details: Participant Flow refers to the Full Analysis Set. First Period started after Baseline (Week 0 to Week 8).
Groups:
- Levetiracetam: * First Period (4 weeks Up-titration and 10 weeks Evaluation): Dry syrup 50 %, 20 mg/kg/day or 1000 mg/day, 40 mg/kg/day or 2000 mg/day, 60 mg/kg/day or 3000 mg/day, twice daily administration Per Os (PO) for 14 weeks.
  * Second Period: Dry syrup 50 % or tablets (250 mg and 500 mg strengths), 20 to 60 mg/kg/day or 1000 to 3000 mg/day, twice daily administration Per Os (PO) until indication granted.
  * Withdrawal Period (6 weeks): Patients on the dose at 60 mg/kg/day or 3000 mg/day will be decreased to 40 mg/kg/day or 2000 mg/day for first 2 weeks and then to 20 mg/kg/day or 1000 mg/day for 2 additional weeks. For patients on the dose at 40 mg/kg/day or 2000 mg/day, the dosage will be decreased to 20 mg/kg/day or 1000 mg/day for 2 weeks and then the treatment with LEV will be stopped.
Period: 1st Period (From Week 8 to Week 22)
Arm/Group | Levetiracetam
Started | 73
Completed | 62 (62 subjects completed the First Period, but 7 of these subjects did not enter the Second Period.)
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 1
Period: 2nd Period (Week 22 to the End of Study)
Arm/Group | Levetiracetam
Started | 55 (7 subjects who completed Period 1 did not enter the Second Period.)
Completed | 35
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 9
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS). FAS includes all subjects taking at least one dose of study medication.
Arm/Group | Levetiracetam
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 41
Region of Enrollment [Number; unit: participants]
  Japan | 73
Age Categorical [Number; unit: participants]
  >=4 - <8 years | 22
  >=8 - <12 years | 22
  >=12 - <16 years | 29
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 32.43 (13.20)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 134.55 (20.69)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram / meter^2 (kg/m^2)] | 17.15 (2.99)
Hospitalization Status [Number; unit: participants]
  Yes | 0
  No | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Partial Seizure Frequency Per Week Over the 14-weeks Treatment Period
Description: The change in partial seizure frequency from Baseline (B) over the Treatment Period (T) is given as a percentage reduction computed as:
  (B values- T values) / B values x 100.
  Positive values in percent reduction mean that the value decreased from Baseline during the first 14-week Period.
  Frequency per week of partial seizures = (Total number of partial seizures in a certain Period/number of observation days in the Period) x 7.
  Partial seizures can be classified into:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: From Baseline (Week 0-8) to the 14-weeks Treatment Period (First Period: 4 weeks Up-titration (Week 8-12) and 10 weeks Evaluation (Week 12-22)); Week 0-22
Population: Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Percent reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 73
Percent reduction | 43.21 [26.19 to 52.14]

2. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs) During the Second Period (up to Three Years Until the Time of Approval Granted)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with the pharmaceutical product. Incidence of treatment-emergent AEs is reported by the percentage of subjects with at least one treatment-emergent AE.
Time Frame: During the second Period from Visit 8 (Week 22) to the end of the Follow-up Period (up to three years until the time of approval granted)
Population: Full Analysis Set (FAS).
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 55
percentage of participants | 98.2

3. Secondary Outcome: Change From Baseline in Partial Seizure Frequency Per Week Over the 10-week Evaluation Period
Description: The change in partial seizure frequency from Baseline (B) over the Evaluation Period (E) is given as a percentage reduction computed as:
  (B values- E values) / B values x 100. Positive values in percent reduction mean that the value decreased from Baseline to the 10-week Evaluation Period.
  Frequency per week of partial seizures = (Total number of partial seizures in a certain Period/number of observation days in the Period) x 7.
  Partial seizures can be classified into:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: From Baseline (Week 0-8) to the 10-weeks Evaluation Period (Part of the first Period: Week 12 to Week 22)
Population: Of the 73 subjects in the FAS, 68 subjects had available data at Baseline and during the Evaluation Period.
Measure: Median (95% Confidence Interval); unit: Percent reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 68
Percent reduction | 39.02 [26.67 to 52.07]

4. Secondary Outcome: Partial Seizure Frequency Per Week Over the 14-weeks Treatment Period
Description: The seizure frequency per week was calculated as:
  Frequency per week of partial seizures = (Total number of partial seizures in the Treatment Period/number of days for observation in the Treatment Period) x 7. Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: 14-weeks Treatment Period (First Period: 4 weeks Up-titration (Week 8-12) and 10 weeks Evaluation (Week 12-22))
Population: Full Analysis Set (FAS). Only subjects having values unequal to zero over Baseline and values equal to or greater than zero over Treatment Period are included.
Measure: Median (Inter-Quartile Range); unit: Seizures per week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 73
Seizures per week | 3.92 [0.93 to 17.08]

5. Secondary Outcome: Partial Seizure Frequency Per Week Over the 10-weeks Evaluation Period
Description: The seizure frequency per week was calculated as:
  Frequency per week of partial seizures = (Total number of partial seizures in the Evaluation Period/number of days for observation in the Evaluation Period) x 7. Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: 10-weeks Evaluation Period (Part of the first Period: Week 12 to Week 22)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Seizures per week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 68
Seizures per week | 3.90 [0.86 to 17.26]

6. Secondary Outcome: Percentage of Partial Seizures 50 % Responders Over the 14-weeks Treatment Period
Description: 50 % responders are those subjects which have a 50 % or more reduction in the frequency of partial seizures from Baseline to the Treatment Period. The results show the percentage of participants that are 50 % responders.
  Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: 14-weeks Treatment Period (First Period: 4 weeks Up-titration (Week 8-12) and 10 weeks Evaluation (Week 12-22))
Population: Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 73
percentage of participants | 38.4 [27.2 to 50.5]

7. Secondary Outcome: Percentage of Partial Seizures 50 % Responders Over the 10-weeks Evaluation Period
Description: 50 % responders are those subjects which have a 50 % or more reduction in the frequency of partial seizures from Baseline to the Evaluation Period. The results show the percentage of participants that are 50 % responders.
  Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: 10-weeks Evaluation Period (Part of the first Period: Week 12 to Week 22)
Population: Of the 73 subjects in the FAS, 68 subjects had available data over the Evaluation Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 68
percentage of participants | 38.2 [26.7 to 50.8]

8. Secondary Outcome: Number of Seizure-free Subjects Over the 14-weeks Treatment Period
Description: Seizure-free means not having a seizure of type I (Partial seizure).
  Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to secondarily generalized seizures.
Time Frame: 14-weeks Treatment Period (First Period: 4 weeks Up-titration (Week 8-12) and 10 weeks Evaluation (Week 12-22))
Population: Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 73
participants | 2

9. Secondary Outcome: Number of Seizure-free Subjects Over the 10-weeks Evaluation Period
Description: as for outcome 8
Time Frame: 10-weeks Evaluation Period (Part of the first Period: Week 12 to Week 22)
Population: Of the 73 subjects in the FAS, 68 subjects had available data over the Evaluation Period.
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 68
participants | 3

10. Secondary Outcome: Incidence of Treatment-emergent Adverse Drug Reactions (ADRs) During the Second Period (up to Three Years Until the Time of Approval Granted)
Description: An Adverse Drug Reaction (ADR) is an Adverse Event for which a causal relationship between the product and the occurrence is suspected. Incidence of ADRs is reported by the number of subjects with at least one ADR.
Time Frame: as for outcome 2
Population: Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 55
participants | 15

11. Secondary Outcome: Change From Baseline in Partial Seizure Frequency Per Week for the Second Period (up to Three Years From Informed Consent Until the Time of Approval Granted)
Description: The outcome was also calculated for each 3-month Period but here only the result for the total Second Evaluation Period (Second Period without following 6-weeks Withdrawal Period for withdrawers) is presented.
  Change in partial seizure frequency from Baseline (B) over Second Evaluation Period (E) is given as a percentage reduction computed as:
  (B values- E values) / B values x 100. Positive values in percent reduction show a decrease from Baseline. Frequency per week of partial seizures = (Total number of partial seizures in a certain Period/number of observation days in the Period) x 7.
Time Frame: From Baseline (Week 0-8) until the time of approval granted (up to three years from date of informed consent (Week 0); without 6-weeks Withdrawal Period)
Population: Full Analysis Set (FAS).
Measure: Median (Inter-Quartile Range); unit: Percent reduction
Arm/Group | Levetiracetam
Number analyzed (Participants) | 55
Percent reduction | 41.32 [15.37 to 82.40]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole study from Baseline (Visit 2) over the complete First Period (14 weeks plus up to 6-week Down-titration and Follow-up) and the Second Period (Week 22 to the end of study).
Description: AEs refer to the Full Analysis Set (FAS). FAS includes all subjects which received at least one dose of study medication.
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 8/73
Other Adverse Events (participants affected / at risk) | 66/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=73)
Strabismus (Eye disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Acetonaemic vomiting (Gastrointestinal disorders) | 1 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=73)
Conjunctivitis (Eye disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (16)
Nausea (Gastrointestinal disorders) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 6 (7)
Dental Caries (Gastrointestinal disorders) | 5 (11)
Pyrexia (General disorders) | 17 (32)
Irritability (General disorders) | 4 (4)
Nasopharyngitis (Infections and infestations) | 54 (205)
Influenza (Infections and infestations) | 20 (24)
Upper respiratory tract infection (Infections and infestations) | 12 (37)
Gastroenteritis (Infections and infestations) | 7 (13)
Impetigo (Infections and infestations) | 4 (4)
Pharyngitis (Infections and infestations) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 8 (11)
Excoriation (Injury, poisoning and procedural complications) | 6 (8)
Wound (Injury, poisoning and procedural complications) | 5 (10)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (21)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Somnolence (Nervous system disorders) | 34 (48)
Headache (Nervous system disorders) | 10 (20)
Convulsion (Nervous system disorders) | 7 (8)
Agitation (Psychiatric disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 6 (6)
Heat rash (Skin and subcutaneous tissue disorders) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days